CLINICAL TRIAL: NCT00283920
Title: PET Imaging of Brain Peripheral Type Benzodiazepine Receptors
Brief Title: PET Imaging of Brain Peripheral Benzodiazepine Receptors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060073; 06-M-0073
Record Dates: First submitted 2006-01-29; First posted 2006-01-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-02

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics; Compartmental Analysis; Distribution Volume; Identitiability; Healthy Volunteer; HV
MeSH Terms: interventions — Carbon-11

INTERVENTIONS:
Drug: [(11)C] PBR28

SUMMARY:
This study will use positron emission tomography (PET) and magnetic resonance imaging (MRI) to measure peripheral benzodiazepine receptors (PBRs) in the brain. PBRs were initially found in peripheral organs such as kidneys, endocrine glands and lungs, but later studies identified PBRs in the CNS. PBRs can be a marker to detect nervous system inflammation. Development of a test to image PBRs may improve the management of brain disorders such as multiple sclerosis, Alzheimer's disease, Parkinson's disease, and others in which inflammation is involved in progression of the disease.

Healthy volunteers from 18 to 40 years old may be eligible for this study. Candidates are screened with tests that may include some or all of the following: diagnostic interview; ratings of mood, anxiety, functioning, and other parameters; neuropsychological testing; physical examination; electrocardiogram; blood and urine tests; and personal, social and family histories.

Participants undergo the following procedures:

* Evaluation: Subjects provide a medical history, including detailed questions about their psychological health, and have a physical examination and blood and urine tests.
* PET scanning: PET uses small amounts of a radioactive chemical called a tracer that "labels" active areas of the brain. The tracer used in this study is [11C]PBR28. For the procedure, the subject lies on the scanner bed. A special mask is fitted to the head and attached to the bed to help keep the head still during the scan so the images will be clear. A brief scan is done just before the radioactive tracer is injected to provide measures of the brain that will help to precisely calculate information from subsequent scans. After the tracer is injected through a catheter (plastic tube) placed in the arm, pictures are taken for 2 to 3 hours, during which the subject lies still on the scanner bed. Subjects return to the clinic the following day for more blood and urine sample collections.
* MRI: The MRI scan is done within 1 year of the PET scan (either before or after the PET). MRI uses magnetic fields and radio waves to produce images of the brain. The patient lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. He or she can communicate with the staff at all times during the procedure.

DETAILED DESCRIPTION:
The peripheral benzodiazepine receptor (PBR) is distinct from central benzodiazepine receptors associated with GABA(A) receptors. Although PBR was initially identified in peripheral organs such as kidneys, endocrine glands and lungs, later studies identified PBR in the central nervous system. In normal conditions, PBR is expressed in low levels in some neurons and glial cells. PBR can be a clinically useful marker to detect neuroinflammation because activated microglial cells in inflammatory areas express much greater levels of PBR than in microglial cells in resting conditions.

PBR has been imaged with positron emission tomography (PET) using [(11)C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195). However, this classical ligand provides only low levels of specific signals and is not sensitive to detect changes occurred in vivo. Recently we developed a new ligand, N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine [(11)C]PBR28, which showed much greater specific signals than [(11)C]PK11195 in non-human primates. In the present protocol, we plan to perform a kinetic brain imaging study in healthy human subjects to measure PBR in brain regions with [(11)C]PBR28. Successful development of a PET ligand to image PBR will have a strong impact on clinical management of brain disorders with inflammation such as multiple sclerosis and ischemia and neurodegenerative disorders such as Alzheimer's and Parkinson's disease where inflammation is involved in the disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All subjects must be healthy and aged 18-65 years.

EXCLUSION CRITERIA:

1. Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.
2. ECG with clinically significant abnormalities. Any existing physical exam and ECG within one year will be reviewed and if none already exists in the chart, these will be obtained and reviewed.
3. Laboratory tests with clinically significant abnormalities.
4. Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits.
5. Pregnancy and breast feeding.
6. Claustrophobia.
7. Presence of ferromagnetic metal in the body or heart pacemaker.
8. Positive HIV test.
9. A history of brain disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-01-26; Study Completion 2007-10-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anholt RR, Pedersen PL, De Souza EB, Snyder SH. The peripheral-type benzodiazepine receptor. Localization to the mitochondrial outer membrane. J Biol Chem. 1986 Jan 15;261(2):576-83. PMID 3001071